CLINICAL TRIAL: NCT04283279
Title: Balance and Mobility in Older Adults With Hearing Impairment
Brief Title: Exercise to Improve Balance in Older Adults With Hearing Impairment - a Proof-of-concept Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Western Norway University of Applied Sciences (Other)
Collaborators: Haukeland University Hospital (Other); University of Dublin, Trinity College (Other)
Responsible Party: Principal Investigator, Bård Bogen, Associate professor, Western Norway University of Applied Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2019/FO243016
Record Dates: First submitted 2019-12-22; First posted 2020-02-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Hearing Loss; Gait, Unsteady; Balance; Distorted; Old Age; Debility
MeSH Terms: conditions — Hearing Loss; Gait Disorders, Neurologic; Frailty | interventions — Exergaming

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual reality exercise (Experimental): 20 participants will be randomised to this arm
  Interventions: Other: Virtual reality exercise
- Vestibular rehabilitation exercise (Experimental): 20 participants will be randomised to this arm
  Interventions: Other: Vestibular rehabilitation exercise
- Control (Other): 20 participants will be randomised to this arm
  Interventions: Other: Control

INTERVENTIONS:
Other: Virtual reality exercise — Participants will do exercises in a virtual environment, solving tasks that require cognitive efforts and motor/balance efforts. The virtual environment/tasks will be delivered through a head-mounted display ("goggles"). Difficulty will progress from standing/sitting, to walking on a treadmill. The environments that will be used will be both over-the-counter environments, as well as in-house designed environments.
  Arms: Virtual reality exercise
Other: Vestibular rehabilitation exercise — Vestibular rehabilitation exercises focus on head and eyes movements, as well as whole-body movements. The aim is to facilitate the use of other sensory organs than the vestibular organs, which will also be relevant to persons who are not receiving sufficient sensory information from the auditory system. The exercises will progress as tolerated, under careful supervision of trained therapists.
  Arms: Vestibular rehabilitation exercise
Other: Control — Participants will not be randomised to either of the exercise interventions, but will be adviced to stay active
  Arms: Control

SUMMARY:
Hearing impairment is common in older adults, and recent research points to associations between hearing impairment and balance/mobility. The association may be due to more attentional resources being used to compensate for the sensory loss, with less resources available for maintaining balance. The aim of this projects is therefore to investigate whether an exercise program with focus on motor-cognitive tasks is feasible for older adults with hearing impairment. The study is meant as a proof-of-concept study, where trialling will be evaluated, and results will be used to inform the design of a larger and adequately powered study.

DETAILED DESCRIPTION:
Study design:

This is an experimental (exercise) study with follow-ups three and twelve months after exercise completion.

Participants:

Participants will be recruited from two instances:

* "Praksisnett", which is a collaboration between GPs and researchers in Bergen, Norway, where GPs recruit potential participants to research projects.
* The Ear, Nose, Throat department at Haukeland University Hospital (Bergen), who provide service to older adults with hearing impairment. The aim is to include 60 patients into three intervention arms: i) virtual reality exercises, ii) vestibular rehabilitation exercises and usual care

Intervention arms:

* Virtual reality exercises: Participants will exercise in virtual environments twice weekly. The choice of environments/tasks will be individualized, and progress from sitting/standing exercises, to doing exercises while walking on a treadmill. The aim is to perform cognitive and motor tasks simultanously.
* Vestibular rehabilitation exercises: This is an exercise approach that has been used in clinical groups, such as patients with vestibular disorders and traumatic brain injury. The aim is to perform movements/exercises where the participant is exposed gradually to movements that may be provocative for the vestibular system.

The exercises will be done in a movement lab at Western Norway University of Applied Sciences. Participants will be randomised to either of the three intervention arms using a computerized procedure. Neither participants, testers or deliverers of the intervention will be blinded. Testers and intervention deliverers will be physiotherapists, students enrolled in a master program in clinical physiotherapy and bachelor students in physiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Hearing threshold above 30 dB

Exclusion Criteria:

* Inability to give informed consent,
* Inability to speak Scandinavian languages or English
* Diseases with severe motor impairments (such as mb Parkinsons)

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Short physical performance battery | Measured as change from baseline/before intervention, to after intervention (six weeks after baseline), to three months after intervention and to 12 months after intervention
  Test of balance and mobility, with three tasks (walking, standing balance, sit-to-stand), scores from 0-12.

SECONDARY OUTCOMES:
Standing balance - posturography | Measured as change from baseline/before intervention, to after intervention (six weeks after baseline), to three months after intervention and to 12 months after intervention
  Body sway measured on a balance platform, with eyes open/closed and on a firm/compliant surface
Walking balance | Measured as change from baseline/before intervention, to after intervention (six weeks after baseline), to three months after intervention and to 12 months after intervention
  Participants will walk across an electronic walkway that registers steps, for analysis of gait steadiness
The World Health Organisation Disability Assessment Schedule (WHODAS) | Measured as change from baseline/before intervention, to after intervention (six weeks after baseline), to three months after intervention and to 12 months after intervention
  Questionnaire that registers disability across several domains. Possible score range is 0-144, where lower values indicate less disability

OTHER OUTCOMES:
Activity monitoring | Measured as change from baseline/before intervention to after intervention (6 weeks after baseline)
  Participants will wear sensors over 4 days, registering activity in their own environments
Dizziness Handicap Inventory | Measured at baseline/before intervention and after intervention (6 weeks after baseline)
  25 item-questionnaire that registers limitations due to dizziness. Possible scores range from 0-100, and higher scores indicate more dizziness-related handicap.